CLINICAL TRIAL: NCT06289998
Title: Phase IIa Clinical Trial of Tamibarotene in Patients With Autosomal Dominant Polycystic Kidney Disease
Brief Title: Study of Tamibarotene in Patients With ADPKD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rege Nephro Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RP014-01
Record Dates: First submitted 2024-02-18; First posted 2024-03-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Keywords: Autosomal dominant polycystic kidney disease
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — tamibarotene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tamibarotene Group (Active Comparator)
  Interventions: Drug: Tamibarotene
- Placebo Group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tamibarotene — Subjects are administrated to tamibarotene 4 mg in daily for 52 weeks.
  Arms: Tamibarotene Group
Drug: Placebo — Subjects are administrated to placebo in daily for 52 weeks.
  Arms: Placebo Group

SUMMARY:
Clinical trial of tamibarotene in patients with Autosomal Dominant Polycystic Kidney Disease

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as ADPKD by modified Pei-Ravine
* eGFR(CKD-EPI) is equal to or greater than 60 mL/min/1.73m^2
* Patients who are judged to be hard to treat with tolvaptan or who do not wish to be treated with tolvaptan, at the time of obtaining consent
* Patients with systolic blood pressure below 140 mmHg and diastolic blood pressure below 90 mmHg. For patients receiving angiotensin-converting enzyme inhibitors or angiotensin II receptor antagonists, the dose must be constant for at least 6 weeks before obtaining informed consent

Exclusion Criteria:

* Women who are pregnant or may be pregnant
* Nursing mother
* Females with childbearing potential or male subjects with a fertile partner who is unable to use contraception for the following periods:

  1. Female: From informed consent to 2 years after the last administration of the study drug
  2. Male: From informed consent to 6 months after the last administration of the study drug
* Patients within 12 weeks from the last dose of a drug that affects renal cysts, such as tolvaptan, to the first dose of the study drug
* Patients with complications of intracranial aneurysm, malignant tumor, uncontrolled diabetes, osteoporosis, uncontrolled dyslipidemia, or abnormal liver function

Ages: 26 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-12-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in TKV from baseline | 52 Week after administration of Investigational Product
  TKV

SECONDARY OUTCOMES:
Changes in TLV from baseline | 52 Week after administration of Investigational Product
  TLV
Changes in eGFR from baseline | 52 Week after administration of Investigational Product
  eGFR
Incidence of adverse events | 1 year
  Safety

CONTACTS AND LOCATIONS:
Locations (8):
- Japan (8):
  - Kurume University Hospital, Kurume, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - Toranomon Hospital Kajigaya, Kawasaki, Kanagawa
  - Kyoto University Hospital, Kyoto, Kyoto
  - Juntendo University School of Medicine Juntendo Hospital, Bunkyo-ku, Tokyo
  - Toranomon Hospital, Minato-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjukuku, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039